CLINICAL TRIAL: NCT03016572
Title: PASS (Promote Access to Stop Suicide): A Randomized Controlled Trial Comparing Enhanced Treatment as Usual, Crisis Center Follow up and Wraparound Services for Youth at Risk for Suicide
Brief Title: Promote Access to Stop Suicide: Comparison of Follow up Services for Youth at Risk for Suicide
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Tatiana Falcone, MD, Tatiana Falcone M.D., The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-886
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Suicide; Depressive Disorder, Major; Anxiety Disorders; Suicidal Ideation; Suicidal Impulses
Keywords: Suicide; Adolescent; Intervention; Crisis; Follow-Up
MeSH Terms: conditions — Suicide; Depressive Disorder, Major; Anxiety Disorders; Suicidal Ideation | interventions — Standard of Care; Crisis Intervention

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Treatment As Usual (E-TAU) (Experimental): The patient will be referred for regular (Standard of Care) outpatient psychiatry/ psychology services or continue with the services that they were receiving prior to admission. They will be followed up by calling patient families at 3 months (post their initial appointment) and at 12 months. They will also have 1 research visit at 6 months (with Dr. Falcone), which they will schedule during their 3 month follow-up call; the Suicide Ideation Questionnaire (SIQ) will be administered. The patients assigned to this group will also be receiving 10 caring follow-up post cards at the following weeks and months (post-discharge from the inpatient unit): 2 weeks, 4 weeks, 6 weeks, 8 weeks, 3 months, 5 months, 7 months, 9 months, 12 months, and on the patient's birthday.
  Interventions: Behavioral: Standard of Care
- TAU + Crisis Center (CC) Follow Up (Experimental): Frontline Services will be administering (at least 9) crisis intervention phone calls to the patients; more calls will be made if they feel it is necessary for the safety and health of the patient. Follow up calls will ask the patient questions about following up in the future, whether they have had thoughts about suicide, whether they are in imminent danger of suicide by the end of the call, and whether the patient is stable. At the end of the call, the patient will be asked to rate their suicidality on a scale of 1 to 10.
  Interventions: Behavioral: Standard of Care; Behavioral: Crisis Intervention
- TAU + CC Follow Up + Wraparound Services (Experimental): This group will be linked with a care coordinator through Tapestry services. Wraparound is an intensive, individualized care coordination and treatment planning process that involves all of the important people in a child's life to work together to make the child successful in school, at home and in the community.
  Interventions: Behavioral: Standard of Care; Behavioral: Crisis Intervention; Behavioral: Wraparound Services

INTERVENTIONS:
Behavioral: Standard of Care — Follow-Up Calls, Questionnaires
Behavioral: Crisis Intervention — Frontline Services will be administering follow up phone calls for participants of the study, recently discharged from the emergency room.
  Arms: TAU + CC Follow Up + Wraparound Services; TAU + Crisis Center (CC) Follow Up
Behavioral: Wraparound Services — Tapestry will be assigning case management services for participants randomized into the third arm of the study.
  Arms: TAU + CC Follow Up + Wraparound Services

SUMMARY:
This research study is designed to answer specific questions about new ways to provide services for youth at-risk of suicide.

DETAILED DESCRIPTION:
The proposed project will be able to provide services to high-risk youth in Ohio. This randomized controlled trial for youth discharged from inpatient psychiatric hospital will be able to determine what combination of services is best suited to reduce subsequent suicide attempts and re-hospitalization.

All youth (ages 10-18), that fit the inclusion criteria, will be recruited from the inpatient unit at Fairview Youth Inpatient Unit. Patients will be consented, enrolled, and assigned to group by the Research Coordinator working at the unit. The Methodologist/ Statistician will generate a random allocation sequence using random number generator and communicate group assignment to the Research Coordinator. There will not be any restriction on randomization. The PI will be blinded to all group assignments.

The clinical research tools and screens that will be administered in this study include: Columbia-Suicide Severity Rating Scale (C-SSRS), The Suicidal Ideation Questionnaire (SIQ), The Adverse Childhood Experiences (ACEs), Ohio Scales, Children's Global Assessment Scale (CGAS), Clinical Global Impressions (CGI-I).

The participants of the study will be seen by the child psychiatrist (Dr. Varkula) and the research coordinator at the initial appointment, and a 6 month follow-up (Dr. Falcone). The C-SSRS and the SIQ will be administered at the initial appointment and the follow-up appointment. The study's research coordinator will be regulating the 3 month phone call and scheduling the 6 month up visit and administering the Ohio Scales questionnaire with the parents and/ or guardians of the child. There will also be a 12 month follow-up phone call conducted by the research coordinator. During this time, the information for the C-SSRS questionnaire, the SIQ, the Ohio Scales (for both the parent and the child), the CGI-I, and the CGAS will be administered.

ELIGIBILITY:
Inclusion Criteria:

* All patients (ages 10-18 years) admitted to the Cleveland Clinic Inpatient Child and Adolescent psychiatry unit after a suicide ideation, behavior, or attempt.
* This can be defined by any intentional, nonfatal self-injury, regardless of medical lethality, will be consider a suicide attempt if intent to die was indicated.
* Signed consent by the adult patient (18 years) or by a first-degree relative or a guardian (for children) at the time of enrollment in the study, and assent by the children as soon as is feasible.

Exclusion Criteria:

* Patients with a known history of autistic spectrum disorder, non-verbal patients and moderate or severe mental retardation (IQ less than 70 and those patients in special education full time), patients with substance dependency and patients with schizophrenia.
* Patients who are enrolled in case management will also be excluded from the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Frequency of repeat suicide attempts in adolescents. | up to 12 months post-discharge
  Frequency of repeat suicide attempts during the 12 month follow up

SECONDARY OUTCOMES:
Frequency of readmissions after a suicide attempt in adolescents. | up to 12 months post-discharge
  Frequency of readmissions after a suicide attempt in adolescents
Relation between service type and frequency of repeat suicide attempts in adolescents. | up to 12 months post-discharge
  Comparing the frequency of repeat suicide attempts in adolescents among the 3 service type treatment arms.
Relation between service type and frequency of readmissions after a suicide attempt in adolescents. | up to 12 months post-discharge
  Comparing the frequency of readmissions after a suicide attempt in adolescents among the 3 service type treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Falcone, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Fairview Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brent DA, Oquendo M, Birmaher B, Greenhill L, Kolko D, Stanley B, Zelazny J, Brodsky B, Firinciogullari S, Ellis SP, Mann JJ. Peripubertal suicide attempts in offspring of suicide attempters with siblings concordant for suicidal behavior. Am J Psychiatry. 2003 Aug;160(8):1486-93. doi: 10.1176/appi.ajp.160.8.1486. PMID 12900312
- [Background] Gould MS, Greenberg T, Velting DM, Shaffer D. Youth suicide risk and preventive interventions: a review of the past 10 years. J Am Acad Child Adolesc Psychiatry. 2003 Apr;42(4):386-405. doi: 10.1097/01.CHI.0000046821.95464.CF. PMID 12649626
- [Background] Nock MK, Green JG, Hwang I, McLaughlin KA, Sampson NA, Zaslavsky AM, Kessler RC. Prevalence, correlates, and treatment of lifetime suicidal behavior among adolescents: results from the National Comorbidity Survey Replication Adolescent Supplement. JAMA Psychiatry. 2013 Mar;70(3):300-10. doi: 10.1001/2013.jamapsychiatry.55. PMID 23303463
- [Background] Torio CM, Encinosa W, Berdahl T, McCormick MC, Simpson LA. Annual report on health care for children and youth in the United States: national estimates of cost, utilization and expenditures for children with mental health conditions. Acad Pediatr. 2015 Jan-Feb;15(1):19-35. doi: 10.1016/j.acap.2014.07.007. Epub 2014 Nov 13. PMID 25444653
- [Background] Gould MS, Kalafat J, Harrismunfakh JL, Kleinman M. An evaluation of crisis hotline outcomes. Part 2: Suicidal callers. Suicide Life Threat Behav. 2007 Jun;37(3):338-52. doi: 10.1521/suli.2007.37.3.338. PMID 17579545
- [Background] Busch KA, Fawcett J, Jacobs DG. Clinical correlates of inpatient suicide. J Clin Psychiatry. 2003 Jan;64(1):14-9. doi: 10.4088/jcp.v64n0105. PMID 12590618